CLINICAL TRIAL: NCT05767086
Title: Comparison of Cetrorelix, Medroxyprogesterone Acetate and Dydrogesterone for Preventing Premature Ovulation in Ovarian Stimulation Cycles
Brief Title: Comparison of 3 Different Protocols for Preventing Premature Ovulation in Ovarian Stimulation Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30.01.2023-E.94828
Record Dates: First submitted 2023-02-27; First posted 2023-03-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Infertility
Keywords: ovulation induction; IVF
MeSH Terms: conditions — Infertility | interventions — cetrorelix; Medroxyprogesterone Acetate; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gonadotropin-releasing hormone (GnRH) antagonist (Experimental): Cetrotide® (0.25 mg, MerckSerono Pharmaceuticals, Darmstadt, Germany)
  Interventions: Drug: Gonadotropin releasing hormone antagonist (Cetrotide)
- Medroxyprogesterone acetate (Experimental): Tarlusal® (5 mg, Deva Pharma, Istanbul, Turkey)
  Interventions: Drug: Medroxyprogesterone Acetate (Tarlusal)
- Dydrogesterone (Experimental): Duphaston® (10mg, Abbott Laboratories, Chicago, Illinois, ABD)
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Gonadotropin releasing hormone antagonist (Cetrotide) — clinical pregnancy rates
  Other Names: Cetrotide
  Arms: Gonadotropin-releasing hormone (GnRH) antagonist
Drug: Medroxyprogesterone Acetate (Tarlusal) — clinical pregnancy rates
  Other Names: Tarlusal
  Arms: Medroxyprogesterone acetate
Drug: Dydrogesterone — clinical pregnancy rates
  Other Names: Duphaston (Duphaston)
  Arms: Dydrogesterone

SUMMARY:
The aim of study is to evaluate the results of three different protocols for prevention of premature ovulation in ovarian stimulation cycles. All patients that undergo IVF cycles are randomly divided into three groups. The first group is cetrorelix, the second group is medroxyprogesterone acetate and the third group is dydrogesterone.

DETAILED DESCRIPTION:
Approximately %10-15 of couples of reproductive age have infertility issues. Ovulation induction and in vitro fertilization (IVF) are the main treatments for infertility. With ovarian stimulation (OS), the efficiency of IVF has been increased by collecting more than one oocytes and thus providing more embryos. Multifollicular growth in OS may cause an increase in sex steroids and an early LH peak, thus premature ovulation. Pituitary suppression with certain drugs has been used to prevent premature ovulation.. Among these drugs, it has been observed that GnRH agonists can cause down-regulation, hypo-estrogenic symptoms, ovarian cyst formation and Ovarian Hyperstimulation Syndrome (OHSS), while antagonists may have side effects such as low oocyte count and high cycle cancellation. The use of progesterone preparations as an alternative to these drugs recently gained ground.

Data including age, BMI, the duration of infertility, the type of infertility, antral follicle count, serum day 3 FSH level, Serum anti-Müllerian hormone level, total gonadotropin dose, stimulation time, pituitary suppression starting day, duration of pituitary suppression, premature ovulation, number of total oocyte count, the number of total M2, the number of PN , the number of Day 5 blast, number of transferred embryos, endometrial thickness on the day of transfer will be recorded. When the follicle size reaches 13-14 mm, patients will be randomized into 3 groups. Group 1 (Cetrorelix: n=99, 0.25 mg/day subcutaneously), Group 2 (Medroxyprogesterone Acetate: n=99, 2x5mg/day orally) and Group 3 (Dydrogesterone: n=99, 3x10 mg/day orally). Human chorionic gonadotropin (hCG) will be used for trigger when at least 2 follicles' diameter reaches 17-18mm for ovulation. Thirty-six hours after the hCG injection, the patient's oocytes will be collected. During 2-5 days of embryo culture, embryo quality will be determined according to D.Gardner criteria (1999). Embryos will be frozen as blast on the 5th day and transferred to the frozen cycle to be planned within the next month. Clinical pregnancy rates will be recorded by performing a blood test for on the 12th day after the procedure.

The aim of this study is to evaluate the results of three different protocols for prevention of premature ovulation in ovarian stimulation cycles. All patients undergo IVF cycles are randomly divided in to three groups. The first group is cetrorelix, the second group is medroxyprogesterone acetate and the third group is dydrogesterone.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-38 years who applied to the infertility clinic
* BMI<25 kg/m2
* AMH>1 ng/mL

Exclusion Criteria:

* Adenomyosis
* Endometriosis
* Untreated uterine pathology
* Hormonal therapy in the last 3 months
* Contraindication for ovulation stimulation
* BMI>25 kg/m2
* AMH<1 ng/mL

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 297 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 4-5 weeks after IVF
  fetal heartbeat by transvaginal ultrasound

SECONDARY OUTCOMES:
Rate of ongoing pregnancy | Months 3
  Ongoing pregnancy rates 3 months after IVF

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ata B, Capuzzo M, Turkgeldi E, Yildiz S, La Marca A. Progestins for pituitary suppression during ovarian stimulation for ART: a comprehensive and systematic review including meta-analyses. Hum Reprod Update. 2021 Jan 4;27(1):48-66. doi: 10.1093/humupd/dmaa040. PMID 33016316
- [Background] Yildiz S, Turkgeldi E, Angun B, Eraslan A, Urman B, Ata B. Comparison of a novel flexible progestin primed ovarian stimulation protocol and the flexible gonadotropin-releasing hormone antagonist protocol for assisted reproductive technology. Fertil Steril. 2019 Oct;112(4):677-683. doi: 10.1016/j.fertnstert.2019.06.009. Epub 2019 Jul 29. PMID 31371053
- [Background] Alexandru P, Cekic SG, Yildiz S, Turkgeldi E, Ata B. Progestins versus GnRH analogues for pituitary suppression during ovarian stimulation for assisted reproductive technology: a systematic review and meta-analysis. Reprod Biomed Online. 2020 Jun;40(6):894-903. doi: 10.1016/j.rbmo.2020.01.027. Epub 2020 Feb 5. PMID 32327297
- [Background] Yang L, Luo K, Lu G, Lin G, Gong F. Euploidy rates among preimplantation genetic testing for aneuploidy cycles with oral dydrogesterone primed ovarian stimulation or GnRH antagonist protocol. Reprod Biomed Online. 2022 Oct;45(4):721-726. doi: 10.1016/j.rbmo.2022.03.003. Epub 2022 Mar 8. PMID 35989167
- [Background] La Marca A, Capuzzo M, Sacchi S, Imbrogno MG, Spinella F, Varricchio MT, Minasi MG, Greco P, Fiorentino F, Greco E. Comparison of euploidy rates of blastocysts in women treated with progestins or GnRH antagonist to prevent the luteinizing hormone surge during ovarian stimulation. Hum Reprod. 2020 Jun 1;35(6):1325-1331. doi: 10.1093/humrep/deaa068. PMID 32395749
- [Result] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417